CLINICAL TRIAL: NCT00435851
Title: Medico-Economic Comparison of Four Strategies of Radioiodine Ablation in Thyroid Carcinoma Patients - Estimabl
Brief Title: Medico-Economic Comparison of Four Strategies of Radioiodine Ablation in Thyroid Carcinoma Patients
Acronym: Estimabl
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Estimabl; CSET 1216
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

INTERVENTIONS:
Drug: Thyrogen, thyroid hormone withdrawal, iode 131

SUMMARY:
In France, 3,700 new cases of thyroid cancer are diagnosed each year. Differentiated thyroid carcinoma represents more than 90% of all thyroid cancers; and has a 10-year survival of 90-95% of patients. This favorable prognosis is the result of an effective primary therapy, which consists of a total thyroidectomy that is followed by radio-iodine ablation with 3,7GBq (100mCi) in case of significant risk of persistent disease. Few centers investigated the possibility to administer lower doses of 131I (1GBq, 30 mCi), in order to limit the potential long-term adverse complications for patients and to respond to radioprotection rules for family members and medical staff.

Radio-iodine ablation requires TSH stimulation, which was historically achieved by thyroid hormone withdrawal for 3 to 5 weeks. During this period, patients suffered from symptoms of hypothyroidism. The recombinant human TSH (rhTSH, Thyrogen®, Genzyme Therapeutics, Cambridge, USA) was approved in Europe in 2005 as an alternative stimulation procedure to withdrawal during ablation. It allows patients to remain euthyroid on thyroid hormone therapy (that needs not to be withdrawn). However, this a costly drug (800 € per patient), whose economic efficiency needs to be checked.

DETAILED DESCRIPTION:
This is a multicentric, randomized, controlled, open-label phase III clinical trial involving 26 French centers. It aims at comparing four strategies of management of postoperative radioiodine ablation, each strategy combining a method of TSH stimulation (thyroid hormone withdrawal or rhTSH (Thyrogen®, Genzyme)) and an activity of 131I (low-dose (1GBq, 30 mCi) or high-dose (3,7GBq, 100 mCi)).

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* Newly diagnosed differentiated papillary or follicular thyroid carcinoma who underwent total thyroidectomy between 30 and 60 days before randomization and treated by LT4 for at least one month.
* Patients are all staged pT1<1cm N1 or pT1>1cm N0 N1 Nx or pT2 N0
* The performance status is 0 or 1.
* All patients will provide written consent to participate.

Exclusion Criteria :

* partial thyroidectomy
* patients treated by LT4 less than one month
* time from thyroidectomy superior to 60 days at randomization
* patients with Hurtle cancer or aggressive histology
* Patients staged pT1<1cm N0 or T2 N1 or T3 or T4 or M1
* patients for which the use of rhTSH is required for medical reasons
* patients with major concurrent medical disorder (cardiac, renal, liver, respiratory)
* patients with other malignancies (exception for in situ cervix uterine cancer, baso cellular skin cancer or breast cancer in remission for at least 2 years)
* patients with recent history of drugs affecting thyroid function, including iodine containing medications or radiocontrast agents
* patients with recent history of 131I whole body scan
* pregant women or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950
Dates: Start 2007-02

PRIMARY OUTCOMES:
the rate of successful postoperative thyroid ablation

SECONDARY OUTCOMES:
the rate of long-term complications
specific toxicities
management costs (hospitalization, diagnosis tests and sick leave)
quality of life and utility

CONTACTS AND LOCATIONS:
Overall Officials: Martin SCHLUMBERGER, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Schlumberger M, Leboulleux S, Catargi B, Deandreis D, Zerdoud S, Bardet S, Rusu D, Godbert Y, Buffet C, Schvartz C, Vera P, Morel O, Benisvy D, Bournaud C, Toubert ME, Kelly A, Benhamou E, Borget I. Outcome after ablation in patients with low-risk thyroid cancer (ESTIMABL1): 5-year follow-up results of a randomised, phase 3, equivalence trial. Lancet Diabetes Endocrinol. 2018 Aug;6(8):618-626. doi: 10.1016/S2213-8587(18)30113-X. Epub 2018 May 26. PMID 29807824
- [Derived] Schlumberger M, Catargi B, Borget I, Deandreis D, Zerdoud S, Bridji B, Bardet S, Leenhardt L, Bastie D, Schvartz C, Vera P, Morel O, Benisvy D, Bournaud C, Bonichon F, Dejax C, Toubert ME, Leboulleux S, Ricard M, Benhamou E; Tumeurs de la Thyroide Refractaires Network for the Essai Stimulation Ablation Equivalence Trial. Strategies of radioiodine ablation in patients with low-risk thyroid cancer. N Engl J Med. 2012 May 3;366(18):1663-73. doi: 10.1056/NEJMoa1108586. PMID 22551127